CLINICAL TRIAL: NCT06012578
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Ascending Dose and Food Effect Study to Evaluate Safety, Tolerability, Pharmacokinetics and Food Effect of ISM5411 in Healthy Subjects
Brief Title: Study Evaluating ISM5411 Administered Orally to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InSilico Medicine Hong Kong Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ISM5411-101
Record Dates: First submitted 2023-08-17; First posted 2023-08-25 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ISM5411 (Experimental)
  Interventions: Drug: ISM5411
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISM5411 — Investigational Drug
  Arms: ISM5411
Drug: Placebo — ISM5411 Matching Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about ISM5411 in healthy subjects. The primary objective is to evaluate the safety and tolerability of single and multiple oral doses of ISM5411 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have signed the informed consent form (ICF) prior to the study, fully understand the content, procedures and possible adverse reactions of the study, and are able to complete the study in accordance with the protocol requirements.
2. Subjects (including their partners) who have no plan to become pregnant and voluntarily use effective contraception as described in section 8.1 from screening to 3 months after the last dose.
3. Male and female subjects aged 18-55 years (inclusive).
4. Body weight ≥50 kg for males and ≥45 kg for females, with a body mass index (BMI = weight (kg)/height2 (m2)) of 18 ~ 32 kg/m2 (inclusive).

Exclusion Criteria:

1. Allergy to the IP or any of its ingredients, or allergic constitution (allergy to more than 1 drugs and food).
2. History of dysphagia or any gastrointestinal surgery (appendicectomy and cholecystectomy are excluded) or disease that affects drug absorption and/or elimination.
3. Presence of clinically relevant diseases evidenced by clinical findings, which are making implementation of the protocol or interpretation of the study results difficult, or that would put the subject at risk by participating in the study in the opinion of the investigator, including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immunological, psychiatric or cardiovascular and cerebrovascular diseases).
4. Presence of abnormal and clinically significant medical history, physical examination, vital signs, 12-lead ECG, clinical laboratory tests, abdominal color Doppler ultrasound, or other investigations at screening (Repeat testing will be allowed by the investigator discretion).
5. Positive human immunodeficiency virus antibody (HIV-Ab), hepatitis B surface antigen (HBsAg) and hepatitis C antibody (HCV-Ab) in the viral serology testing at screening.
6. Smoking > 5 cigarettes or an equivalent amount of tobacco per day, or consuming ≥ 14 units of alcohol per week (1 unit of alcohol ≈ 25 mL of spirits/100 mL of wine/285 mL of beer) within 1 months prior to screening or unwilling to abstain from smoking or drinking during the study.
7. Subjects who are positive for urine drug testing at screening or Day-1, or have a history of drug abuse or narcotic use in the past five years (Repeat testing will be allowed by the investigator discretion).
8. Subjects who have donated blood or lost a significant amount of blood (>400 mL) within 1 months prior to screening, or who plan to donate blood during the study or within 1 month after the end of the study.
9. Subjects who have undergone major surgical procedures (major visceral, organ, or bone surgeries) that may affect the study in the judgment of the investigator within 3 months prior to screening, or who intend to have such procedures during the study.
10. Intolerance to vein puncture, or presence of a history of blood phobia or trypanophobia.
11. Use of any prescription drugs within 14 days prior to the admission. Use of counter medication / vitamins / supplements within 7 days prior to admission (with the exception of contraception, occasional paracetamol, and standard dose of multivitamins).
12. Subjects who have receipt of any study drug or participated in any medical device clinical studies within 1 month (or 5 half-lives, whichever is longer) prior to screening.
13. Vaccination with any live or attenuated vaccine within 1 month prior to screening.
14. Any acute disease or acute attack of any chronic disease within 28 days prior to screening.
15. Consumption of any caffeinated food or beverages (such as coffee, strong tea, cola, chocolate, etc.), xanthine-rich food (such as anchovies, sardines, bovine liver, bovine kidney, etc.), food that induces or inhibits liver metabolizing enzymes (such as dragon fruits, mango, grapefruit, pomegranate, etc.) and beverages made thereof, or food or beverages containing alcohol, or presence of other factors that may affect the absorption, distribution, metabolism or excretion of the drug (such as strenuous exercise) within 48 hours prior to IP.
16. Female subjects who are in lactation or positive for serum pregnancy test during the screening period or study course.
17. Subjects who, in the judgment of the investigator, are not suitable for participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) after single or multiple doses of ISM5411. | Up to 7 days after last dose.
  The number of participants with treatment related AEs as assessed by CTCAE v5.0. will be monitored.
Number of participants with clinically significant changes in vital signs | Up to 7 days after last dose.
  The number of participants with clinically significant changes in vital signs will be monitored based on the assessment of blood pressure, heart rate, respiration and body temperature before and after administration.
Number of participants with clinically significant changes in in chemistry laboratory values | Up to 7 days after last dose
  The number of participants with clinically significant changes in blood routine, blood biochemistry, urine routine, coagulation function, etc. will be monitored before and after administration.
Number of participants with clinically significant changes in 12-lead Electrocardiogram (ECG) readings | Up to 7 days after last dose
  The number of participants with clinically significant changes in 12-lead Electrocardiogram (ECG) readings will be monitored based on changes in cardiovascular system function (change in QTC parameters) as a criterion of safety and tolerability variables.
Number of participants with clinically significant changes in physical examinations | Up to 7 days after last dose
  Complete physical examination should include the head and face, skin system, lymph nodes, eyes, ears, nose and throat, mouth, respiratory system, cardiovascular system, abdomen, musculoskeletal system, nervous system and mental status.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Time at which the maximum plasma concentration occurred (tmax) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Area under the plasma concentration-time curve from time zero to time with last measurable concentration t (AUC0-t) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Elimination rate constant (λz) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Elimination half-life (t1/2) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Apparent volume of distribution (Vz/F) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Apparent total plasma clearance (CL/F) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Mean residence time (MRT) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Renal clearance rate (CLR) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Accumulative excretion (Ae) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Fractional excretion (fe) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.
Relative bioavailability (fed/fasted) of ISM5411 | Day 1 through Day 17
  To evaluate the pharmacokinetics (PK) characteristics of ISM5411 in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No